CLINICAL TRIAL: NCT02197988
Title: Efficacy and Safety of Transversus Abdominis Plane Blocks Versus Thoracic Epidural Anesthesia in Patients Undergoing Major Abdominal Resections: A Prospective, Randomized Controlled Trial
Brief Title: TAP Versus Thoracic Epidural in Major Abdominal Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-218
Record Dates: First submitted 2014-05-13; First posted 2014-07-23 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Malignant Neoplasm of Abdomen; Surgery
Keywords: Surgery; Abdominal; Epidural Anesthesia; Transversus Abdominis Plane Block; TAP block
MeSH Terms: interventions — Fentanyl; Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transversus Abdominis Plane Block (Active Comparator): Transversus Abdominis Plane Block Exparel 1.33% (20ml Volume)
  Interventions: Drug: Exparel 1.33% (20ml Volume)
- Thoracic Epidural Anesthesia (Active Comparator): Thoracic Epidural Anesthesia 0.125% bupivicaine with 2 mcg/ml Fentanyl
  Interventions: Drug: 0.125% bupivicaine with 2 mcg/ml Fentanyl.

INTERVENTIONS:
Drug: Exparel 1.33% (20ml Volume) — Transversus Abdominis Plane Block
  Other Names: TAP Block; Transversus Abdominis Plane Block
  Arms: Transversus Abdominis Plane Block
Drug: 0.125% bupivicaine with 2 mcg/ml Fentanyl. — Thoracic Epidural Anesthesia
  Other Names: Epidural; Thoracic Epidural Anesthesia
  Arms: Thoracic Epidural Anesthesia

SUMMARY:
The purpose of this study is to compare two standard methods of pain control management used at Spectrum Health for patients undergoing major surgery. The two methods being compared are the thoracic epidural and the TAP block. The thoracic epidural method involves medication being given through a patient's back and the TAP block involves medication being given through a patient's abdomen (belly). The investigators will compare side effects experienced by the patients that take part in this study, including a change in blood pressure, as well as the patients' opinions about their pain management experience after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical profiles of two currently acceptable analgesia techniques in terms of incidence of hypotension with subsequent fluid administration and pain control by evaluation of both objective and subjective data. The investigators will also compare any additional hospital costs associated with side effect management related to either analgesia method.

This study is a prospective, randomized, open-label trial. Patients who agree to participate and satisfy the inclusion/exclusion criteria will be randomized at the time of enrollment into one of two groups (thoracic epidural or TAP block) using a randomization tool created for the study.

Patients will undergo their scheduled surgery and receive the analgesic method to which they have been randomized. Both methods (thoracic epidural or TAP block) are performed routinely at Spectrum Health and are considered routine care.

Data collected will include medical history and demographics from the patient's medical record. Intraoperative data will include length of surgery, estimated surgical blood loss, complications, blood pressure and medication requirements. Postoperative data will include episodes of hypotension (defined as a systolic BP < 90), fluid requirement in first 24 hours and first 72 hours, pain scores, narcotic usage, return to bowel function (as defined by flatus), time to tolerating a soft or regular diet, and complications. Data will also be collected via a survey each study patient will complete for study purposes only.

ELIGIBILITY:
Inclusion Criteria:

* All patients male or female >18 years old who are scheduled to undergo a major abdominal surgery. Abdominal procedures include, but are not limited to: pancreaticoduodenectomies, distal pancreatectomies, bowel resection, liver resection, esophagectomies, heated intraperitoneal chemotherapy, retroperitoneal excisions and large genitourinary procedures
* Patients determined by their surgeon as medically able to receive a thoracic epidural or a TAP block interchangeably after consideration of both procedures
* Patient agrees to participate in this study and provides informed consent

Exclusion criteria:

* Surgical cases combined with thoracic surgeries
* Surgical cases where the abdominal operation is performed laparoscopically
* Patients that have allergies to lidocaine, bupivacaine, levobupivacaine or hydromorphone
* Patients that are on anticoagulation or antiplatelet medications at time of surgery other than aspirin
* Surgical cases that typically do not require a regional block in addition to general anesthesia (e.g., cutaneous operations)
* Adults unable to provide informed consent
* Children
* Pregnant women
* Prisoners
* Non-English speaking subjects
* Any other medical condition including mental illness or substance abuse deemed by the investigator to be likely to interfere with a subject's ability to provide informed consent, cooperate and take part in this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Hypotension | First 24-72 hours postoperatively
  The incidence of systolic blood pressure less than 90 mmHg and fluid requirements

SECONDARY OUTCOMES:
Patient satisfaction relative to pain control and amount of additional narcotic usage | Post operative day two during hospitalization
  A short patient survey during the postoperative period which will collect information on pain management.

OTHER OUTCOMES:
Cost Evaluation | Postoperative hospitalization an expected average of 6 months
  Evaluate costs incurred relative to adverse side effect management and pain management related to either the TAP block or thoracic epidural.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Chung, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518
- [Background] Torup H, Mitchell AU, Breindahl T, Hansen EG, Rosenberg J, Moller AM. Potentially toxic concentrations in blood of total ropivacaine after bilateral transversus abdominis plane blocks; a pharmacokinetic study. Eur J Anaesthesiol. 2012 May;29(5):235-8. doi: 10.1097/EJA.0b013e328350b0d5. PMID 22450529
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Conaghan P, Maxwell-Armstrong C, Bedforth N, Gornall C, Baxendale B, Hong LL, Carty HM, Acheson AG. Efficacy of transversus abdominis plane blocks in laparoscopic colorectal resections. Surg Endosc. 2010 Oct;24(10):2480-4. doi: 10.1007/s00464-010-0989-y. Epub 2010 Apr 8. PMID 20376492
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Taylor R Jr, Pergolizzi JV, Sinclair A, Raffa RB, Aldington D, Plavin S, Apfel CC. Transversus abdominis block: clinical uses, side effects, and future perspectives. Pain Pract. 2013 Apr;13(4):332-44. doi: 10.1111/j.1533-2500.2012.00595.x. Epub 2013 Feb 13. PMID 22967210
- [Background] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327
- [Background] Holte K, Foss NB, Svensen C, Lund C, Madsen JL, Kehlet H. Epidural anesthesia, hypotension, and changes in intravascular volume. Anesthesiology. 2004 Feb;100(2):281-6. doi: 10.1097/00000542-200402000-00016. PMID 14739801
- [Background] Hilton AK, Pellegrino VA, Scheinkestel CD. Avoiding common problems associated with intravenous fluid therapy. Med J Aust. 2008 Nov 3;189(9):509-13. doi: 10.5694/j.1326-5377.2008.tb02147.x. PMID 18976194
- [Background] Niraj G, Kelkar A, Jeyapalan I, Graff-Baker P, Williams O, Darbar A, Maheshwaran A, Powell R. Comparison of analgesic efficacy of subcostal transversus abdominis plane blocks with epidural analgesia following upper abdominal surgery. Anaesthesia. 2011 Jun;66(6):465-71. doi: 10.1111/j.1365-2044.2011.06700.x. Epub 2011 Apr 4. PMID 21457153